CLINICAL TRIAL: NCT07404176
Title: Terbium-161 DOTATATE in Metastatic Neuroendocrine Tumors: Assessment of Safety and Efficacy
Brief Title: Study to Assess the Safety and Effectiveness of Novel Radiopharmaceutical Terbium-161 DOTATATE in Metastatic Neuroendocrine Tumors
Acronym: TENET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Ameya Puranik, Professor, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMCIEC4940; REF/2026/01/120894 (Other: Clinical Trial Registry of India)
Record Dates: First submitted 2026-01-23; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Neuroendocrine Neoplasms (Tumours); Neuroendocrine Tumors; Metastatic Neuroendocrine Tumors
Keywords: Terbium 161; metastatic NET; DOTATATE
MeSH Terms: conditions — Neoplasms; Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: Simon 2-stage
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Terbium 161 DOTATATE PRRT (Experimental): Peptide Receptor Radionuclide Therapy with 7.4 GBq of Terbium 161 DOTATATE administered every 6-8 weeks
  Interventions: Drug: Terbium 161

INTERVENTIONS:
Drug: Terbium 161 — Auger-emitter Peptide Receptor Radionuclide Therapy

SUMMARY:
Gastro-enteropancreatic Neuro-endocrine tumors (GEP-NETs) are rare slow-growing cancers which commonly involve the abdominal organs like liver, stomach, intestines and pancreas. Their incidence has been documented to have increased over the last decade, thus resulting in treatment options being developed to treat these cancers. These cancers spread commonly to the liver, followed by lungs, bones and other sites. Depending on the extent of disease seen on scan, treatment is planned. Patients are advised Peptide Receptor Radionuclide Therapy (PRRT), which is the current standard of treatment for metastatic GEP-NETs. Radio-isotopes labeled to octreotide analogs bind to somatostatin receptors on surface of cancer cells and deliver radiation to the cancer cells when injected into the body. Lu-177 (Lutetium-177) is one such radioisotope which has been used for tagging to the octreotide and is known as Lu-177 DOTATATE PRRT, which is now routinely used in clinical practice. Terbium-161 is another radioisotope which can be labeled to octreotide and used for PRRT. It has advantages over Lu-177 such that it specifically reaches the tumor sites and does not affect the surrounding normal cells, due to its higher penetrating capacity and shorter range of travel. This will benefit patients as the effectiveness of PRRT will be higher with lesser side effects. However, the investigators can only do this by performing a study. Response to treatment can be evaluated by performing scans and side effects, if any can be studied by performing blood tests.

DETAILED DESCRIPTION:
Targeted radionuclide therapy (TRT) is a nuclear medicine technique that uses radiopharmaceuticals (RPs) with high affinity to receptors or antigens on the surface of tumor cells to achieve a therapeutic effect. TRT causes less collateral damage than external beam radiotherapy (EBRT) because the RPs are selectively taken up by tumors and their metastases, delivering high doses of radiation to cancer cells and minimizing doses to normal tissues.NETTER-1 and 2 trials have already established PRRT (Peptide Receptor Radionuclide Therapy) with Lutetium-177 (Lu-177) DOTATATE as first line TRT in metastatic well-differentiated gastro-enteropancreatic neuroendocrine tumors(GEP-NETs).

While Lu-177 as a radioisotope is safe and indigenously produced by BARC, the recent global shortage of this isotope has led to development of Terbium-161 (Tb-161). Terbium-161 belongs to the same family of Lanthanides as Lu-177 and offers the same physical characteristics.

The superiority of Tb-161 over Lu-177 evolves from its basic property of emission of Auger electrons (AE).(4) Most important characteristics of radioisotopes in Nuclear Medicine or Radiation Oncology are linear energy transfer and range; which are determinants of cell-damage to the target cell and normal cell, respectively. Compared to beta-emissions (as in Lu-177), AEs are most lethal to cancer cells when emitted near the cell nucleus and especially when incorporated into DNA. AEs cause DNA damage both directly and indirectly via water radiolysis. AEs can also kill targeted cancer cells by damaging the cell membrane and producing more targeted and lethal effects. Moreover, the important point is that since the range of delivery of this energy is relatively shorter as compared to beta-emitters, hence there is negligible bystander and crossfire effect, thereby causing no damage to surrounding cells.

Monte-Carlo simulations: Larauze et al assessed absorbed doses from simulations performed with CELLDOSE, which is a homemade Monte Carlo track-structure code for simulating the transport of electrons in water, based on differential and total interaction cross sections describing the elastic scattering, electronic excitation, and ionization. Absorbed doses to cell nuclei and cell membranes (with an intranuclear radionuclide location, only nuclear absorbed doses were assessed) were assessed. In this tumor cluster model, when all cells were targeted, and depending on the location of the radionuclide, Tb-161 delivered a 2- to 3-fold higher nuclear absorbed doses than Lu-177 but also 2- to 6-fold higher absorbed doses to cell membranes. Interaction of ionizing radiation with the cell membrane induces sphingomyelin hydrolysis to ceramide, initiating apoptosis.

Spoormans et al performed cellular dosimetry to quantify the absorbed dose to the cell nucleus and compared dose-response curves to evaluate differences in relative biological effectiveness in vitro, between Tb-161 and Lu-177. (7) Tb-161-DOTATATE and delivered a 3.6 times higher dose to the nucleus, respectively, than their Lu-177-labeled counterparts on saturated receptor binding. This increased nucleus-absorbed dose was mainly due to the additional emission of internal conversion electrons by Tb-161.

Verberg et al did a comparative dosimetric analysis of Lu-177 DOTATATE and Tb-161 DOTATATE by calculating the radiation absorbed dose to tumor as well as non-target organs of normal biodistribution, on adult human phantom models. The substitution of Lu-177 with Tb-161 results in an increase in the delivered dose per unit of activity to tumour tissue by 40% (in a 10 g tumour: 2.9 Gy/GBq and 4.1 Gy/GBq, respectively) as well as to dose-limiting non-target tissue (kidneys: 39%(0.73 Gy/GBq and 1.01 Gy/GBq, respectively), bone marrow: 42% (0.04 Gy/GBq and 0.06 Gy/GBq, respectively)

First-In-Human Studies: After qualifying through the cell survival and dosimetry studies, Baum et al used Tb-161 DOTATATE in 2 patients, one with paraganglioma and other with metastatic neuroendocrine tumor, both of whom were refractory to Lu-177 DOTATATE therapy. Patients formally consent to receive this treatment and Tb-161 DOTATATE was administered following the standard PRRT protocol. Post therapy SPECT/CT images were acquired which showed tracer localisation at the desired tumor locations. No adverse events and no changes in vital parameters were observed or reported by the patient during, immediately after or at follow-up review of the patient after administration of Tb-161-DOTATATE. According to the Common Terminology Criteria for Adverse Events, there were no clinically significant changes in the relevant laboratory values (hematological, renal, and hepatic panel) at the subsequent follow up of the patient after administration of Tb-161-DOTATATE.

Dept of Nuclear Medicine, TMH and ACTREC has already obtained approval from Atomic Energy Regulatory Board (AERB), and has treated 2 patients of metastatic NET on compassionate basis with Tb-161 DOTATATE, who were refractory to Lu-177 DOTATATE.

The investigators therefore would like to study the safety and efficacy of Tb-161 DOTATATE in patients in metastatic NET who have shown disease progression after treatment with Lu-177 DOTATATE PRRT.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age greater than 18 years
* Histopathological diagnosis of well-differentiated GEP-NET
* Positive Ga-68-DOTANOC PET/CT, Krennings score >/=3
* Locally advanced/inoperable disease or metastatic disease
* Patient who have shown disease progression with Lu-177 DOTATATE PRRT
* Karnofsky performance-status score of at least 60 or ECOG performance status </=2
* Life expectancy greater than 6 months

Exclusion Criteria:

* Serum creatinine level of more than 1.6 mg/dl or a creatinine clearance of less than 50 ml/min
* Hemoglobin level of less than 8.0 g per deciliter
* Red blood cell count less than 300,000/cubic millimeter
* White cell count of less than 2000 per cubic millimeter
* Platelet count of less than 75,000 per cubic millimetre
* Total bilirubin level of more than 3 times the upper limit of the normal range
* Serum albumin level > 3.0 g/dl
* Pregnancy and Lactation
* Patients with concurrent malignancies

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Disease control rate | 4-6 weeks
  Disease control rate will be measured as a primary endpoint. It is percentage of patients achieving complete or partial response or stable disease on Ga-68 DOTATATE PET/CT. Response assessment will be done using RECIST 1.1 for solid tumors. Non-PD (non-disease progression) after one session of Tb-161 therapy will be eligible for the second session. Patients showing CR with no residual measurable disease will not undergo a second session of therapy. Patients with PD after 1 cycle of Tb-161 DOTATATE therapy will not continue in the study

SECONDARY OUTCOMES:
Quality of Life assessment | Before therapy, at 4 weeks and 8 weeks after each therapy session.
  Clinical and Quality of Life Assessment using EORTC QLQ C30
Safety Assessment | 2 weeks, 4 weeks and 6 weeks after each therapy
  At each visit, the investigator will evaluate the subject to determine whether any AEs have occurred. CBC, LFT, RFT, Serum electrolytes will be done at 2 weeks, 4 weeks and 6 weeks after each therapy. AEs may be directly observed, reported spontaneously by the subject or by questioning the subject at each study visit. All laboratory values will be evaluated by the Investigator as to clinical significance. All post-baseline abnormal laboratory values considered clinically significant by the Investigator will be recorded as an AE. The NCI Common Terminology Criteria for Adverse Events version 5 (NCI CTCAE v5.0) will be used to classify and grade the intensity of adverse events during and after each treatment cycle. CTCAE will be used to grade all events regardless of attribution, in order to ensure objective reporting, and in order to report trial data according to accepted international guidelines. The highest grade of each observed toxicity will be recorded.
Quality of Life assessment using QLQ-GI.NET21 questionnaire | Before therapy, at 4 weeks and 8 weeks after each therapy session.
  Clinical and Quality of Life Assessment using EORTC QLQ-GI.NET21

CONTACTS AND LOCATIONS:
Overall Officials: Ameya Puranik, DNB, Principal Investigator — Tata Memorial Hospital, Mumbai
Locations (2):
- India (2):
  - Tata Memorial Hospital, Mumbai, India, Mumbai, Maharashtra
  - Advanced Centre for Treatment, Research and Education in Cancer (ACTREC), Navi Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided
Not approved by institutional ethics committee

REFERENCES:
- [Background] Baum RP, Singh A, Kulkarni HR, Bernhardt P, Ryden T, Schuchardt C, Gracheva N, Grundler PV, Koster U, Muller D, Prohl M, Zeevaart JR, Schibli R, van der Meulen NP, Muller C. First-in-Humans Application of 161Tb: A Feasibility Study Using 161Tb-DOTATOC. J Nucl Med. 2021 Oct;62(10):1391-1397. doi: 10.2967/jnumed.120.258376. Epub 2021 Feb 5. PMID 33547209
- [Background] Verburg FA, de Blois E, Koolen S, Konijnenberg MW. Replacing Lu-177 with Tb-161 in DOTA-TATE and PSMA-617 therapy: potential dosimetric implications for activity selection. EJNMMI Phys. 2023 Nov 10;10(1):69. doi: 10.1186/s40658-023-00589-w. PMID 37947917

DOCUMENTS (1):
  • Study Protocol (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/76/NCT07404176/Prot_000.pdf